CLINICAL TRIAL: NCT04545736
Title: Oral Metformin for Treatment of ABCA4 Retinopathy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200163; 20-EI-0163
Record Dates: First submitted 2020-09-10; First posted 2020-09-11 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10-23

CONDITIONS: ABCA4 Retinopathy; Stargardt Disease; Retinal Dystrophy; Retinal Degeneration
Keywords: Stargardt Disease; Retinal Dystrophy; Retinal Degeneration
MeSH Terms: conditions — Stargardt Disease; Retinal Dystrophies; Retinal Degeneration | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metformin (Experimental): Oral administration of metformin
  Interventions: Drug: Metformin hydrochloride

INTERVENTIONS:
Drug: Metformin hydrochloride — Metformin is commercially produced in immediate and extended release. Participants will receive an immediate release formulation of metformin of 500mg daily at study entry. This dose will be titrated up weekly in 500mg increments to reach a goal of 2000mg daily maximum. Once participants >=17 years of age reach 2000mg metformin immediate release they will switch to an extended-release formulation (1000mg twice a day by mouth). Participants >= 17 years of age that cannot tolerate 2000mg will be permitted to reduce their daily dose to a minimum of 1000mg/day. Because metformin extended release is not FDA-approved for children under the age of 17, participants under 17 will remain on the immediate release formulation. For these participants who remain on standard formulation, the maximum tolerated dose between 1000mg and 2000mg/day will be given.

SUMMARY:
Background:

ABCA4 retinopathy is a genetic disease in which the ABCA4 protein is absent or faulty. It can cause waste material to collect in the eye and may cause cells to die. The cell death can lead to vision loss. Researchers want to see if an oral drug called metformin can help.

Objective:

To see if metformin is safe and possibly helps to slow the rate of ABCA4 retinopathy.

Eligibility:

People age 12 and older who have ABCA4 retinopathy and have problems with their vision.

Design:

Participants will be screened under a separate protocol.

Participants will have a medical and family history. They will complete a questionnaire about their vision and daily activities. They will have a physical exam. They may have blood drawn through a needle in the arm.

Participants will have an eye exam. Their pupils may be dilated with eye drops. Their retina may be photographed.

Participants will have a visual field test. They will sit in front of a large dome and press a button when they see a light within the dome.

Participants will have an electroretinogram. It examines the function of the retina. They will sit in the dark for 30 minutes. Then their eyes will be numbed with eye drops. They will wear contact lenses that can sense signals from the retinas. They will watch flashing lights.

Participants will have optical coherence tomography. This non-invasive procedure makes pictures of the retina.

Participants will have fundus autofluorescence. A bright blue light will be shone into their eye.

Participants will take metformin by mouth for 24 months.

Participants will have study visits every 6 months. Participation will last for at least 36 months....

DETAILED DESCRIPTION:
Study Description:

ABCA4 retinopathy is an autosomal recessive progressive retinal dystrophy that leads to retinal pigment epithelium (RPE) and photoreceptor degeneration, with consequent central visual loss. A treatment that either reduces the rate of lipofuscin accumulation or improves the clearance of lipofuscin in the RPE could potentially slow the degeneration associated with this disease. Metformin hydrochloride is a well-characterized, commonly prescribed oral anti-diabetic medication that acts by suppressing liver gluconeogenesis and increasing peripheral insulin sensitivity.

An additional effect of metformin is to increase macroautophagy via the Mammalian target of rapamycin complex 1 (mTORC1)/AMP-activated Kinase (AMPK) pathway; stimulation of this pathway would be predicted to enable the RPE to more efficiently handle lipofuscin. This suggests an association between metformin use and slowing of retinal degeneration. The objective of this study is to investigate the safety and potential efficacy of oral metformin in slowing the rate of change in photoreceptor degeneration in ABCA4 retinopathy.

Objectives:

The objective of this study is to investigate the safety and potential efficacy of oral metformin in slowing the rate of change in photoreceptor degeneration in ABCA4 retinopathy.

Endpoints:

Primary Endpoint: The difference in growth rate of square-root transformed area of EZ band loss (square-root AreaEZloss), from OCT, between the pre-treatment phase and 24 month metformin treatment phase.

Secondary Endpoints: Proportion of participants with a 30% reduction in growth rate of square-root AreaEZloss during the treatment phase compared to the pre-treatment phase, changes from baseline to Month 24 in Best-Corrected Visual Acuity (BCVA) total letters read, perimetry, and color fundus photography measurements and the change in rate of area of atrophy enlargement between the pre-treatment and 24-month metformin treatment phase.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant must be at least 12 years of age.
2. Participant (or legal guardian) must understand and sign the protocol s informed consent document.
3. Participant must have at least one definite pathogenic or likely pathogenic mutation in ABCA4 and a typical clinical presentation of Stargardt disease and phenotypic presentation of ABCA4 retinopathy in both eyes.
4. Participant must have at least two years of natural history data from at least four data points (a) The separation between any two consecutive data points must be at least six months (b) The most recent data point must be at least 4.5 months and no more than 16 months prior to the baseline visit (c)

   1. Potential participants with three natural history data points may be enrolled to obtain their fourth natural history data point on protocol.
   2. The separation between any two consecutive data points may fall short of 6 months by no more than 45 days; however, the total separation among the data points must allow for at least two years of natural history data.
   3. Potential participants with four or more natural history data points completed off protocol, all of which having occurred more than 16 months prior to the baseline visit, may be enrolled to complete an additional natural history data point on protocol within the required timeframe from the baseline visit.
5. Participant must agree to adhere to Lifestyle Considerations throughout study duration.
6. Any female participant of childbearing potential must have a negative urine pregnancy test at screening and be willing to undergo urine pregnancy tests throughout the study.
7. Any female participant of childbearing potential must:

   * Have had a surgical sterilization OR
   * Completely abstain from intercourse OR
   * Practice at least one form of contraception while actively taking IP on the study and at least one week after IP discontinuation OR
   * Have a partner who had a surgical sterilization OR
   * Have a partner who practices one form of contraception while the female participant is actively taking IP and at least one week after the female participant discontinues IP.

Any male participants must:

* Have had a surgical sterilization OR
* Completely abstain from intercourse OR
* Practice at least one form of contraception while actively taking IP on the study and at least for 3 months after IP discontinuation OR
* Have a partner who had a surgical sterilization OR
* Have a partner who practices one form of contraception while the male participant actively takes IP and at least 3 months after the male participant discontinues IP.

  1. Acceptable forms of surgical sterilization include: vasectomy, hysterectomy, or tubal ligation.
  2. Acceptable methods of contraception include: hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, or barrier methods (diaphragm, condom) with spermicide.

     EXCLUSION CRITERIA:

     An individual who meets any of the following criteria will be excluded from participation in this study:
     1. Participant is actively receiving study IP in another investigational study.
     2. Participant has a condition that would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control) by interfering with the participant s ability to engage in the required protocol evaluation and testing and/or comply with study visits.
     3. Any female participant of childbearing potential that is pregnant or breast-feeding at the time of enrollment or planning to become pregnant during the study.
     4. Participant has definitive pathogenic or likely pathogenic mutations in RDS/peripherin (PRPH2), PROM1, and/or ELOVL4.
     5. Participant has a history of chronic renal impairment as measured in the acute care panel estimated glomerular filtration rate (eGFR)<45 ml/min/1.73 m2) or severe hepatic, pulmonary, or cardiovascular disease (hypoxic state).
     6. Participant is taking any medication that could adversely interact with metformin (e.g., cimetidine, furosemide, nifedipine) and cannot switch to an alternative medication.
     7. Participant is currently taking metformin or participant has taken metformin during the period of natural history data collection that will be used for this study for a cumulative total of more than one month (> 31 days).
     8. Participant has a known hypersensitivity to metformin.
     9. Participant has not stopped taking a glucagon-like peptide 1 (GLP-1) agonist at least two weeks prior to enrollment or is currently taking a GLP-1 agonist.
     10. Participant has a history of chronic lactic acidosis, including diabetic ketoacidosis, with or without coma.
     11. Participant has type 1 diabetes mellitus.
     12. Scarring due to choroidal neovascularization (CNV) is present in either eye.

     QUALIFYING EYE ELIGIBILITY CRITERIA:

     In order to participate in the study, the participant must have at least one qualifying eye that meets all of the inclusion and none of the exclusion criteria listed below.

     Qualifying Eye Inclusion Criteria:

     1. A growth rate of square root AreaEZloss > 0.025 mm/year based on calculation from natural history data.

     Qualifying Eye Exclusion Criteria:

     1. Retinal degeneration has advanced beyond a point where reliable measurement of the integrity of the IS-OS on OCT is possible.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The difference in growth rate of square-root transformed area of EZ band loss (vAreaEZloss) | Pre-treatment, Baseline, Month 24
  The difference in growth rate of vAreaEZloss, from OCT, between the pre-treatment phase and treatment phase.

SECONDARY OUTCOMES:
Proportion of participants with a 30% reduction in growth rate of vAreaEZloss | Pre-treatment, Baseline, Month 24
  Proportion of participants with 30% reduction in growth rate of vAreaEZloss, from OCT, during the treatment phase compared to the pre-treatment phase.
Number and severity of adverse events | ongoing throughout study
  The number and severity of systemic and ocular toxicities, adverse events and infections by severity, type and assessed relatedness to the IP throughout the study period.
Changes in best corrected visual acuity (BCVA) | Baseline, Month 24
  The change in BCVA total letters read from baseline to Month 24.
Change in rate of area of atrophy enlargement | Pre-treatment, Baseline, Month 24
  The difference in rate of region of atrophy measurements from FAF between the pre-treatment phase and treatment phase.
Change in perimetry and color fundus photography measurements | Baseline, Month 24
  The change in perimetry and color fundus photography from baseline to Month 24.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-EI-0163.html